CLINICAL TRIAL: NCT00074854
Title: A Clinical Efficacy Study Of An Oral Tyrosine Kinase Inhibitor Of VEGFR-2 Given In Combination With Chemotherapy (Paclitaxel And Carboplatin) Vs. Chemotherapy Alone For The Treatment Of Advanced Stage Non-Small Cell Lung Cancer.
Brief Title: A Clinical Efficacy Study Of An Oral Tyrosine Kinase Inhibitor Of VEGFR-2 Given In Combination With Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3521002
Record Dates: First submitted 2003-12-22; First posted 2003-12-24 (Estimated); Last update posted 2006-11-09 (Estimated); Status verified 2006-07

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — 3-(4-bromo-2,6-difluorobenzyloxy)-5-(3-(4-pyrrolidin-1-ylbutyl)ureido)isothiazole-4-carboxylic acid amide

INTERVENTIONS:
Drug: CP-547,632

SUMMARY:
The purpose of this study is to determine whether CP-547,632, an oral VEGFR-2 tyrosine kinase inhibitor when given in combination with chemotherapy (carboplatin and paclitaxel) is effective in the treatment of advanced stage non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB (inicluding those with pleural effusion), IV or recurrent non-small cell lung cancer (nsclc).
* Bidimensionally measurable disease >2cm x 1 cm by conventional CT Scan or >1 cm x 1cm by spiral CT Scan.

Exclusion Criteria:

* No tumors in close proximity to major veins or arteries.
* No sanguinous pleural effusion due to disease or pericardial effusion suspicious for disease.
* No evidence or history brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87
Dates: Start 2002-05; Study Completion 2005-03

PRIMARY OUTCOMES:
Statistical estimates used on the Stage 1 data indicated low likely-hood of a positive outcome if the study continued to Stage 2. This provided the basis for discontinuation of the trial.

SECONDARY OUTCOMES:
Given the outcome of the primary objective, analysis of secondary objectives were not formalized.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, San Mateo, California
  - Pfizer Investigational Site, San Pablo, California
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3521002&StudyName=A+Clinical+Efficacy+Study+Of+An+Oral+Tyrosine+Kinase+Inhibitor+Of+VEGFR%2D2+Given+In+Combination+With+Chemotherapy